CLINICAL TRIAL: NCT04298905
Title: Leveraging mHealth to Enable and Adapt Community Health Worker Strategies to Improve TB/HIV Patient Outcomes in South Africa (LEAP-TB-SA) Trial
Brief Title: Leveraging mHealth to Enable and Adapt CHW Strategies to Improve TB/HIV Patient Outcomes in SA
Acronym: LEAP-TB-SA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: University of Witwatersrand, South Africa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00211518
Record Dates: First submitted 2020-03-04; First posted 2020-03-06 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Adherence, Patient; TB; HIV/AIDS; Care Coordination
Keywords: mHealth; community health worker; TB/HIV
MeSH Terms: conditions — Patient Compliance; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Study design overview: LEAP-TB-SA is a pilot randomized controlled trial. There are two arms: mHealth intervention (100) and health education control (100).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Individuals randomized to standard of care will receive a standardized adherence education session and provided with a paper-based diary to track appointments and adherence. Instructions will be provided on the importance of daily adherence in the primary health care facility closest to patients' residence, as per standard of care. Directly observed therapy (DOT) is recommended for all patients at patients' nearest clinic. All patients are seen face-to-face monthly for adherence monitoring, monthly symptom reports and laboratory evaluations per standard of care treatment guidelines. All research participants will also receive a clinic visit quality checklist to ensure completeness of standard of care procedures.
- mHealth intervention (Active Comparator): Individuals randomized to the intervention arm will receive the same standardized adherence education, followed by an orientation session to the study intervention. This orientation will include education on basic smartphone operations and use. The CHW will set up appointment reminders for clinic visits as well as daily adherence reminders for submission of the video DOT sessions and symptom reports. A smartphone capable of downloading apps, receiving short message service (SMS) and access wifi and cellular connectivity will be provided to intervention patients. All patients are seen face-to-face monthly for adherence monitoring, monthly symptom reports and laboratory evaluations per standard of care treatment guidelines. All research participants will also receive a clinic visit quality checklist to ensure completeness of standard of care procedures.
  Interventions: Other: CHW mHealth patient intervention for trigger escalation

INTERVENTIONS:
Other: CHW mHealth patient intervention for trigger escalation — The CHW dashboard is a tablet-based, per-patient summary of the patient intervention. It is this dashboard that identifies a trigger to escalate the adherence intervention. This dashboard is created by receiving information from the patient's smartphone application as well as the National Health Laboratory Service (NHLS) data feed of laboratory results. The monitoring features included in this dashboard:
  1. NHLS laboratory results: Dashboard receives and flags NHLS results for any positive smear or culture (new positive after prior negative results) or detectable viral load (with prior viral suppression)
     1. Triggered, escalating adherence coaching:
     2. Safety monitoring: reports all abnormal laboratory values to provider
  2. Appointment keeping (RETAIN):
     a. Triggered, escalating adherence coaching
  3. vDOT submissions:
     a. Triggered, escalating adherence coaching
  4. Symptom reports:
     1. Triggered, escalating adherence coaching
  Arms: mHealth intervention

SUMMARY:
mHealth solutions designed to support affordable human resources for health, such as community health workers (CHWs), offer the opportunity to reimagine a patient-centered, system-level solution that may radically change care models in low resource settings. The 'leap' of m-health is most potent and practical in settings where desktop-based infrastructure is lacking and hard-wired internet connectivity is unavailable.

Investigators have demonstrated the feasibility of mHealth and human resource solutions in South Africa and shown marked improvements in screening, linkage and treatment initiation as well as supporting patient adherence through video DOT (vDOT) and early identification of treatment related toxicity. Investigators' strategies have evaluated solutions for individual cascade steps through TB and HIV smartphone and tablet-based m-health applications implemented by a CHW. This study combines these individual cascade step approaches into an innovative TB/HIV cascade intervention study entitled, "Leveraging mHealth to enable and adapt community health worker strategies to improve TB/HIV patient outcomes in South Africa (LEAP-TB-SA) Trial."

DETAILED DESCRIPTION:
Mycobacterium tuberculosis (TB) is the leading cause of death for persons living with HIV (PLWH) in South Africa (SA). Estimates suggest that if factoring in immediate lost to follow-up, a mere 52% of TB/HIV co-infected individuals have successful treatment outcomes. Factors contributing to this bleak reality occur throughout the TB/HIV cascade and include: limited capacity for TB screening; delays in linkage or failure to link into care; treatment non-adherence; and long and toxic treatment regimens that lead to disengagement in care. Reducing mortality and improving TB treatment outcomes among PLWH requires system-level, patient-centered interventions that enhance movement along both cascades. Through innovative mobile health (mHealth) approaches, designed to optimize human resources, and create efficiency for all users and engage patients in care, it is possible to reduce system bottlenecks and rapidly improve treatment outcomes.

Studies addressing the TB or HIV care cascades are increasingly common, yet few offer an integrated, sustainable approach to TB/HIV co-infection and, to date, no intervention spans the entire cascade. The TB/HIV care cascade begins with diagnosis of TB in a PLWH or in a person newly diagnosed with both diseases. Patients newly diagnosed with TB and HIV face a burdensome model of care influenced by: a) timing of HIV treatment initiation; b) worsened symptom profiles associated with immune reconstitution syndrome; c) higher pill burden; d) differential adherence challenges; e) and more frequent care visits for directly observed therapy (DOT) and laboratory evaluations. Many, have struggled with adherence to HIV regimen, prior to the TB diagnosis. Data found that 44% of PLWH on anti-retroviral therapy (ART) present with viral suppression to first TB visit, suggesting the need to further intensify adherence interventions in this group.

Hypothesis: The intervention will have fewer composite negative TB outcomes (i.e. treatment failure, loss to follow-up, and death) compared to attention controls.

Primary Aims:

1. to determine the feasibility, acceptability and impact of a mHealth triggered, escalating adherence intervention by community health workers (CHW) to improve rif-resistant (RR)-TB treatment outcomes among PLWH in Kwa-Zulu Natal, Province of South Africa through a pilot randomized controlled trial. H1. the mHealth triggered, escalating adherence intervention by CHW's will improve treatment success for RR-TB and HIV co-infected patients compared to attention control participants.

Secondary Aims:

1. to conduct a time-limited prospective screening cohort of close contacts of persons diagnosed with RR-TB using respondent driven sampling.
2. to evaluate willingness to participate in the trial and determine who screen fails for any reason.
3. to evaluate study process indicators to further refine the behavioral and technological components of the intervention (patient symptom reporting; vDOT submission compliance; CHW adherence coaching sessions; intervention theoretical models; and mHealth application feature enhancements to support care coordination).
4. to characterize the emergence of resistance among patients with non-adherence to RR-TB treatment, by obtaining two additional sputum specimens (i.e., 1) on treatment initiation for all patients and 2) among participants with a 30-day period of less than optimal adherence (defined as <90% of vDOT submissions or patient/provider report non-adherence) and/or treatment failure (defined as positive culture with evidence of additional antimicrobial resistance) to fully characterize resistance patterns through genotypic and phenotypic resistance testing as well as next generation molecular sequencing.
5. to characterize HIV genotypic resistance patterns among participants with a detectable viral load.
6. to determine, retrospectively, the impact of HIV resistance patterns on RR-TB treatment outcomes.
7. to assess stigma throughout the RR-TB care continuum and evaluate whether the level of stigma changes through different phases of treatment.
8. to pilot test the psychometric properties of four novel indicators of intersectional RR- TB-HIV stigma.

ELIGIBILITY:
Inclusion Criteria:

* Any person 18 years of age or older with pulmonary TB
* HIV positive
* Outpatient TB treatment (including short course RR-TB treatment) or admission < 30 days is expected

Exclusion Criteria:

* Unwilling or unable to provide informed consent, including inability to consent in one of the approved languages
* Patients who require hospitalization for TB treatment at treatment initiation
* Extrapulmonary or disseminated TB disease
* Severe clinical presentation: BMI < 18 kg/m2 or a person unable to stand/walk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment success | Up to 12 months
  Treatment success is defined as cure and completion of treatment.
Number of deaths among participants | Up to 12 months
  Number of death (all causes) among participants will be assessed.
Number of participants with treatment failure | Up to 12 months
  Treatment failure is defined as worsening antimicrobial resistance.
Number of participants lost to follow-up | Up to 12 months
  Loss to follow-up is defined as 2 or more consecutive months of missed treatment.

SECONDARY OUTCOMES:
Time to linkage to care | Up to 30 days
  Time (days) to linkage to care for TB.
Time to treatment initiation | Up to 30 days
  Time (days) to treatment initiation for TB.

CONTACTS AND LOCATIONS:
Overall Officials: Jason E Farley, PhD, MPH, Principal Investigator — Johns Hopkins University School of Nursing
Locations (1):
- Kelly Lowensen, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Geneva. Global Tuberculosis Report 2018.; 2018. doi:ISBN 978 92 4 156539 4
- [Background] Naidoo P, Theron G, Rangaka MX, Chihota VN, Vaughan L, Brey ZO, Pillay Y. The South African Tuberculosis Care Cascade: Estimated Losses and Methodological Challenges. J Infect Dis. 2017 Nov 6;216(suppl_7):S702-S713. doi: 10.1093/infdis/jix335. PMID 29117342
- [Background] Seid A, Metaferia Y. Factors associated with treatment delay among newly diagnosed tuberculosis patients in Dessie city and surroundings, Northern Central Ethiopia: a cross-sectional study. BMC Public Health. 2018 Jul 28;18(1):931. doi: 10.1186/s12889-018-5823-9. PMID 30055593
- [Background] Takarinda KC, Harries AD, Nyathi B, Ngwenya M, Mutasa-Apollo T, Sandy C. Tuberculosis treatment delays and associated factors within the Zimbabwe national tuberculosis programme. BMC Public Health. 2015 Jan 29;15:29. doi: 10.1186/s12889-015-1437-7. PMID 25631667
- [Background] Meintjes G, Schoeman H, Morroni C, Wilson D, Maartens G. Patient and provider delay in tuberculosis suspects from communities with a high HIV prevalence in South Africa: a cross-sectional study. BMC Infect Dis. 2008 May 25;8:72. doi: 10.1186/1471-2334-8-72. PMID 18501019
- [Background] Gebremariam MK, Bjune GA, Frich JC. Barriers and facilitators of adherence to TB treatment in patients on concomitant TB and HIV treatment: a qualitative study. BMC Public Health. 2010 Oct 28;10:651. doi: 10.1186/1471-2458-10-651. PMID 21029405
- [Background] Naidoo P, Peltzer K, Louw J, Matseke G, McHunu G, Tutshana B. Predictors of tuberculosis (TB) and antiretroviral (ARV) medication non-adherence in public primary care patients in South Africa: a cross sectional study. BMC Public Health. 2013 Apr 26;13:396. doi: 10.1186/1471-2458-13-396. PMID 23622516
- [Background] Amuha MG, Kutyabami P, Kitutu FE, Odoi-Adome R, Kalyango JN. Non-adherence to anti-TB drugs among TB/HIV co-infected patients in Mbarara Hospital Uganda: prevalence and associated factors. Afr Health Sci. 2009 Aug 1;9 Suppl 1(Suppl 1):S8-15. PMID 20589161
- [Background] Van der Walt M, Lancaster J, Odendaal R, Davis JG, Shean K, Farley J. Serious treatment related adverse drug reactions amongst anti-retroviral naive MDR-TB patients. PLoS One. 2013;8(4):e58817. doi: 10.1371/journal.pone.0058817. Epub 2013 Apr 3. PMID 23573193
- [Background] Farley JE, Ram M, Pan W, Waldman S, Cassell GH, Chaisson RE, Weyer K, Lancaster J, Van der Walt M. Outcomes of multi-drug resistant tuberculosis (MDR-TB) among a cohort of South African patients with high HIV prevalence. PLoS One. 2011;6(7):e20436. doi: 10.1371/journal.pone.0020436. Epub 2011 Jul 22. PMID 21799728
- [Background] Lessells RJ, Swaminathan S, Godfrey-Faussett P. HIV treatment cascade in tuberculosis patients. Curr Opin HIV AIDS. 2015 Nov;10(6):439-46. doi: 10.1097/COH.0000000000000197. PMID 26352390
- [Background] Shapiro AE, van Heerden A, Schaafsma TT, Hughes JP, Baeten JM, van Rooyen H, Tumwesigye E, Celum CL, Barnabas RV. Completion of the tuberculosis care cascade in a community-based HIV linkage-to-care study in South Africa and Uganda. J Int AIDS Soc. 2018 Jan;21(1):e25065. doi: 10.1002/jia2.25065. PMID 29381257
- [Background] Hanrahan CF, Van Rie A. A proposed novel framework for monitoring and evaluation of the cascade of HIV-associated TB care at the health facility level. J Int AIDS Soc. 2017 Apr 20;20(1):21375. doi: 10.7448/IAS.20.01.21375. PMID 28440604
- [Background] Havlir DV, Kendall MA, Ive P, Kumwenda J, Swindells S, Qasba SS, Luetkemeyer AF, Hogg E, Rooney JF, Wu X, Hosseinipour MC, Lalloo U, Veloso VG, Some FF, Kumarasamy N, Padayatchi N, Santos BR, Reid S, Hakim J, Mohapi L, Mugyenyi P, Sanchez J, Lama JR, Pape JW, Sanchez A, Asmelash A, Moko E, Sawe F, Andersen J, Sanne I; AIDS Clinical Trials Group Study A5221. Timing of antiretroviral therapy for HIV-1 infection and tuberculosis. N Engl J Med. 2011 Oct 20;365(16):1482-91. doi: 10.1056/NEJMoa1013607. PMID 22010914
- [Background] Abdool Karim SS, Naidoo K, Grobler A, Padayatchi N, Baxter C, Gray AL, Gengiah T, Gengiah S, Naidoo A, Jithoo N, Nair G, El-Sadr WM, Friedland G, Abdool Karim Q. Integration of antiretroviral therapy with tuberculosis treatment. N Engl J Med. 2011 Oct 20;365(16):1492-501. doi: 10.1056/NEJMoa1014181. PMID 22010915
- [Background] Naidoo K, Yende-Zuma N, Padayatchi N, Naidoo K, Jithoo N, Nair G, Bamber S, Gengiah S, El-Sadr WM, Friedland G, Abdool Karim S. The immune reconstitution inflammatory syndrome after antiretroviral therapy initiation in patients with tuberculosis: findings from the SAPiT trial. Ann Intern Med. 2012 Sep 4;157(5):313-24. doi: 10.7326/0003-4819-157-5-201209040-00004. PMID 22944873
- [Background] Daftary A, Padayatchi N, O'Donnell M. Preferential adherence to antiretroviral therapy over tuberculosis treatment: a qualitative study of drug-resistant TB/HIV co-infected patients in South Africa. Glob Public Health. 2014;9(9):1107-16. doi: 10.1080/17441692.2014.934266. Epub 2014 Jul 18. PMID 25035943
- [Background] Louw J, Peltzer K, Naidoo P, Matseke G, Mchunu G, Tutshana B. Quality of life among tuberculosis (TB), TB retreatment and/or TB-HIV co-infected primary public health care patients in three districts in South Africa. Health Qual Life Outcomes. 2012 Jun 28;10:77. doi: 10.1186/1477-7525-10-77. PMID 22742511
- [Background] Tsui S, Denison JA, Kennedy CE, Chang LW, Koole O, Torpey K, Van Praag E, Farley J, Ford N, Stuart L, Wabwire-Mangen F. Identifying models of HIV care and treatment service delivery in Tanzania, Uganda, and Zambia using cluster analysis and Delphi survey. BMC Health Serv Res. 2017 Dec 6;17(1):811. doi: 10.1186/s12913-017-2772-4. PMID 29207973
- [Background] Gandhi NR, Moll AP, Lalloo U, Pawinski R, Zeller K, Moodley P, Meyer E, Friedland G; Tugela Ferry Care and Research (TFCaRes) Collaboration. Successful integration of tuberculosis and HIV treatment in rural South Africa: the Sizonq'oba study. J Acquir Immune Defic Syndr. 2009 Jan 1;50(1):37-43. doi: 10.1097/QAI.0b013e31818ce6c4. PMID 19295333
- [Background] Abstract: Heidari, Omeid (Johns Hopkins University School of Nursing); Nguyen, Yen ((Johns Hopkins University School of Nursing); Budhathoki, Chakra (Johns Hopkins University School of Nursing); Geiger, Keri (Johns Hopkins University School of Nursing); Stamper, P (Johns Hopkins School of Nursing); Farley, JE (Johns Hopkins University School of Nursing. Evaluating HIV 90-90-90 Targets for Individuals with Drug-Resistant Tuberculosis Treatment in South Africa. 2019.
- [Background] Kelly AM, Smith B, Luo Z, Given B, Wehrwein T, Master I, Farley JE. Discordance between patient and clinician reports of adverse reactions to MDR-TB treatment. Int J Tuberc Lung Dis. 2016 Apr;20(4):442-7. doi: 10.5588/ijtld.15.0318. PMID 26970151
- [Background] Han HR, Kim K, Murphy J, Cudjoe J, Wilson P, Sharps P, Farley JE. Community health worker interventions to promote psychosocial outcomes among people living with HIV-A systematic review. PLoS One. 2018 Apr 24;13(4):e0194928. doi: 10.1371/journal.pone.0194928. eCollection 2018. PMID 29689054
- [Background] Uwimana J, Zarowsky C, Hausler H, Jackson D. Training community care workers to provide comprehensive TB/HIV/PMTCT integrated care in KwaZulu-Natal: lessons learnt. Trop Med Int Health. 2012 Apr;17(4):488-96. doi: 10.1111/j.1365-3156.2011.02951.x. Epub 2012 Feb 1. PMID 22296235
- [Background] Hoffman JA, Cunningham JR, Suleh AJ, Sundsmo A, Dekker D, Vago F, Munly K, Igonya EK, Hunt-Glassman J. Mobile direct observation treatment for tuberculosis patients: a technical feasibility pilot using mobile phones in Nairobi, Kenya. Am J Prev Med. 2010 Jul;39(1):78-80. doi: 10.1016/j.amepre.2010.02.018. Epub 2010 May 26. PMID 20537846
- [Background] Farley JE, McKenzie-White J, Bollinger R, Hong H, Lowensen K, Chang LW, Stamper P, Berrie L, Olsen F, Isherwood L, Ndjeka N, Stevens W. Evaluation of miLINC to shorten time to treatment for rifampicin-resistant Mycobacterium tuberculosis. Int J Tuberc Lung Dis. 2019 Sep 1;23(9):980-988. doi: 10.5588/ijtld.18.0503. PMID 31615604
- [Background] Holzman SB, Zenilman A, Shah M. Advancing Patient-Centered Care in Tuberculosis Management: A Mixed-Methods Appraisal of Video Directly Observed Therapy. Open Forum Infect Dis. 2018 Apr 26;5(4):ofy046. doi: 10.1093/ofid/ofy046. eCollection 2018 Apr. PMID 29732378
- [Background] Fisher JD, Fisher WA, Amico KR, Harman JJ. An information-motivation-behavioral skills model of adherence to antiretroviral therapy. Health Psychol. 2006 Jul;25(4):462-73. doi: 10.1037/0278-6133.25.4.462. PMID 16846321
- [Background] Horvath KJ, Smolenski D, Amico KR. An empirical test of the information-motivation-behavioral skills model of ART adherence in a sample of HIV-positive persons primarily in out-of-HIV-care settings. AIDS Care. 2014 Feb;26(2):142-51. doi: 10.1080/09540121.2013.802283. Epub 2013 Jun 3. PMID 23724908
- [Background] May CR, Cummings A, Girling M, Bracher M, Mair FS, May CM, Murray E, Myall M, Rapley T, Finch T. Using Normalization Process Theory in feasibility studies and process evaluations of complex healthcare interventions: a systematic review. Implement Sci. 2018 Jun 7;13(1):80. doi: 10.1186/s13012-018-0758-1. PMID 29879986
- [Background] Atkins S, Lewin S, Ringsberg KC, Thorson A. Provider experiences of the implementation of a new tuberculosis treatment programme: a qualitative study using the normalisation process model. BMC Health Serv Res. 2011 Oct 17;11:275. doi: 10.1186/1472-6963-11-275. PMID 22004533
- [Background] Farley JE, Ndjeka N, Kelly AM, Whitehouse E, Lachman S, Budhathoki C, Lowensen K, Bergren E, Mabuza H, Mlandu N, van der Walt M. Evaluation of a nurse practitioner-physician task-sharing model for multidrug-resistant tuberculosis in South Africa. PLoS One. 2017 Aug 4;12(8):e0182780. doi: 10.1371/journal.pone.0182780. eCollection 2017. PMID 28783758
- [Background] Farley JE, Kelly AM, Reiser K, Brown M, Kub J, Davis JG, Walshe L, Van der Walt M. Development and evaluation of a pilot nurse case management model to address multidrug-resistant tuberculosis (MDR-TB) and HIV in South Africa. PLoS One. 2014 Nov 18;9(11):e111702. doi: 10.1371/journal.pone.0111702. eCollection 2014. PMID 25405988
- [Background] Usabilit.gov. System Usability Scale (SUS). usability.gov. doi:10.1007/s10339
- [Background] Hong H, Budhathoki C, Farley JE. Increased risk of aminoglycoside-induced hearing loss in MDR-TB patients with HIV coinfection. Int J Tuberc Lung Dis. 2018 Jun 1;22(6):667-674. doi: 10.5588/ijtld.17.0830. PMID 29862952